CLINICAL TRIAL: NCT04564547
Title: A Phase 2b, Randomized, Active-Controlled, Double-Blind, Dose-Ranging Clinical Study to Evaluate a Switch to Islatravir (ISL) and MK-8507 Once-Weekly in Adults With HIV-1 Virologically Suppressed on Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/FTC/TAF) Once-Daily
Brief Title: Dose Ranging, Switch Study of Islatravir (MK-8591) and Ulonivirine (MK-8507) Once-Weekly in Virologically-Suppressed Adults With Human Immunodeficiency Virus Type 1 (HIV-1) [MK-8591-013]
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8591-013; MK-8591-013 (Other: MSD Protocol Number); 2024-511041-19-00 (Registry Identifier: EU CT); U1111-1302-9886 (Registry Identifier: UTN); 2020-003071-18 (EudraCT Number)
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — islatravir; ulonivirine; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In study Part 1 (double-blind treatment period), a double-blinding technique with in-house blinding is used. Ulonivirine, ISL, and BIC/FTC/TAF will be packaged identically relative to their matching placebos so that the blind is maintained. The participant, the investigator, and Sponsor personnel or delegate(s) who are involved in the study intervention administration or clinical evaluation of the participants are unaware of the intervention assignments.
  In the unblinded safety monitoring period, participants, investigators, and Sponsor personnel are unblinded as to the participant's original randomized intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: ISL 20 mg + Ulonivirine 100 mg (Experimental): Participants receive ISL 20 mg + ulonivirine 100 mg once weekly (QW) and placebo to BIC/FTC/TAF once daily (QD). Following study-wide discontinuation of study intervention, participants may have entered the optional unblinded safety monitoring period and received standard of care non-study ART.
  Interventions: Drug: Islatravir; Drug: Ulonivirine; Drug: Placebo to Ulonivirine; Drug: Placebo to BIC/FTC/TAF
- Group 2: ISL 20 mg + Ulonivirine 200 mg (Experimental): Participants receive ISL 20 mg + ulonivirine 200 mg QW and placebo to BIC/FTC/TAF QD. Following study-wide discontinuation of study intervention, participants may have entered the optional unblinded safety monitoring period and received standard of care non-study ART.
  Interventions: Drug: Islatravir; Drug: Ulonivirine; Drug: Placebo to Ulonivirine; Drug: Placebo to BIC/FTC/TAF
- Group 3: ISL 20 mg + Ulonivirine 400 mg (Experimental): Participants receive ISL 20 mg + ulonivirine 400 mg QW and placebo to BIC/FTC/TAF QD. Following study-wide discontinuation of study intervention, participants may have entered the optional unblinded safety monitoring period and received standard of care non-study ART.
  Interventions: Drug: Islatravir; Drug: Ulonivirine; Drug: Placebo to BIC/FTC/TAF
- Group 4: BIC/FTC/TAF (Active Comparator): Participants receive placebo to ISL + placebo to ulonivirine QW and BIC/FTC/TAF 50 mg/200 mg/25 mg QD.
  Interventions: Drug: BIC/FTC/TAF; Drug: Placebo to ISL; Drug: Placebo to Ulonivirine

INTERVENTIONS:
Drug: Islatravir — ISL capsule taken by mouth.
  Other Names: MK-8591
  Arms: Group 1: ISL 20 mg + Ulonivirine 100 mg; Group 2: ISL 20 mg + Ulonivirine 200 mg; Group 3: ISL 20 mg + Ulonivirine 400 mg
Drug: Ulonivirine — Ulonivirine tablet taken by mouth.
  Other Names: MK-8507
  Arms: Group 1: ISL 20 mg + Ulonivirine 100 mg; Group 2: ISL 20 mg + Ulonivirine 200 mg; Group 3: ISL 20 mg + Ulonivirine 400 mg
Drug: BIC/FTC/TAF — BIC/FTC/TAF tablet taken by mouth.
  Other Names: BIKTARVY®
  Arms: Group 4: BIC/FTC/TAF
Drug: Placebo to ISL — Placebo capsule matched to ISL taken by mouth.
  Arms: Group 4: BIC/FTC/TAF
Drug: Placebo to Ulonivirine — Placebo tablet matched to ulonivirine taken by mouth.
  Arms: Group 1: ISL 20 mg + Ulonivirine 100 mg; Group 2: ISL 20 mg + Ulonivirine 200 mg; Group 4: BIC/FTC/TAF
Drug: Placebo to BIC/FTC/TAF — Placebo tablet matched to BIC/FTC/TAF taken by mouth.
  Arms: Group 1: ISL 20 mg + Ulonivirine 100 mg; Group 2: ISL 20 mg + Ulonivirine 200 mg; Group 3: ISL 20 mg + Ulonivirine 400 mg

SUMMARY:
This is a randomized, controlled, double-blind, study to evaluate the safety and tolerability of islatravir (ISL) + ulonivirine based on review of the accumulated safety data, in adult participants with human immunodeficiency virus type 1 (HIV-1) who have been virologically suppressed for ≥6 months on bictegravir/emtricitabine/tenofovir alafenamide (BIC/FTC/TAF) once-daily.

DETAILED DESCRIPTION:
Based on laboratory findings of decreased lymphocyte and CD4+ T-cell counts across the islatravir program and as described in protocol amendment 2 (approved 01-Dec-2021), participants in study Part 1 (double-blind treatment period) were unblinded, discontinued all study interventions, and switched to standard of care non-study antiretroviral (ART) therapy. Participants who received ISL + ulonivirine (Groups 1 to 3) may have then entered into an unblinded safety monitoring period and were monitored for ≥6 months. As specified in protocol amendment 2, study Parts 2 and 3 were no longer planned or initiated for any participant.

ELIGIBILITY:
Inclusion Criteria:

* Is HIV-1 positive with plasma human immunodeficiency virus type 1 (HIV-1) RNA <50 copies/mL at screening
* Has been virologically suppressed on bictegravir/emtricitabine/tenofovir alafenamide (BIC/FTC/TAF) for ≥6 months
* Has a screening CD4+ T-cell count >200 cells/mm^3 (completed by the central laboratory)
* Is male or female, at least 18 years of age, at the time of signing the informed consent
* Female participants are eligible to participate if not pregnant or breastfeeding, and at least one of the following conditions applies:

  * Is not a woman of childbearing potential (WOCBP)
  * Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis)

Exclusion Criteria:

* Has HIV-2 infection
* Has hypersensitivity or other contraindication to any of the components of the study interventions as determined by the investigator
* Has active hepatitis C virus (HCV) coinfection (defined as detectable HCV RNA) or hepatitis B virus (HBV) coinfection (defined as hepatitis B surface antigen [HBsAg]-positive or HBV deoxyribonucleic acid [DNA] positive)
* Has a current (active) diagnosis of acute hepatitis due to any cause
* Has a history of malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or cutaneous Kaposi's sarcoma
* Has a history or current evidence of any condition (including active tuberculosis infection), therapy, laboratory abnormality or other circumstance (including drug or alcohol use or dependence) that might, in the opinion of the investigator, confound the results of the study or interfere with the participant's participation for the full duration of the study
* Is taking or is anticipated to require systemic immunosuppressive therapy, immune modulators, or any prohibited therapies
* Is currently participating in or has participated in a clinical study with an investigational compound or device from 45 days prior to Day 1 through the study treatment period
* Has a documented or known virological resistance to ulonivirine or nucleoside/nucleotide reverse transcriptase inhibitors (NNRTI)
* Is female and expecting to conceive or donate eggs at any time during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (23):
- United States (10):
  - Pueblo Family Physicians ( Site 2702), Phoenix, Arizona
  - Men's Health Foundation ( Site 2710), Los Angeles, California
  - Midway Immunology and Research ( Site 2713), Ft. Pierce, Florida
  - Triple O Research Institute, P.A. ( Site 2712), West Palm Beach, Florida
  - Infectious Disease Specialists Of Atlanta PC ( Site 2704), Decatur, Georgia
  - Chatham County Health Department ( Site 2707), Savannah, Georgia
  - Kansas City CARE Clinic ( Site 2703), Kansas City, Missouri
  - Saint Hope Foundation, Inc. ( Site 2716), Bellaire, Texas
  - Texas Centers for Infectious Disease Associates P.A. ( Site 2709), Fort Worth, Texas
  - DCOL Center for Clinical Research ( Site 2715), Longview, Texas
- France (8):
  - CHU de Toulouse - Hopital Purpan ( Site 2302), Toulouse, Haute-Garonne
  - Hopital Gui de Chauliac. ( Site 2303), Montpellier, Herault
  - CHU Hotel Dieu Nantes ( Site 2310), Nantes, Loire-Atlantique
  - Centre Hospitalier Regional du Orleans ( Site 2304), Orléans, Loiret
  - Hopital Avicenne ( Site 2305), Bobigny, Seine-Saint-Denis
  - Hopital Saint Louis ( Site 2308), Paris
  - Hopital Saint-Antoine ( Site 2307), Paris
  - Pitie Salpetriere University Hospital-Infectious Disease - Tropical Diseases ( Site 2306), Paris, Île-de-France Region
- Switzerland (5):
  - Universitaetsspital Zuerich ( Site 2601), Zuerich, Canton of Aargau
  - Universitaetsspital Basel ( Site 2602), Basel, Canton of Basel-City
  - Inselspital Universitaetsspital Bern ( Site 2603), Bern, Canton of Bern
  - Hopitaux Universitaires de Geneve HUG ( Site 2604), Geneva, Canton of Geneva
  - CHUV (centre hospitalier universitaire vaudois) ( Site 2605), Lausanne, Canton of Vaud

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26181&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As pre-specified in protocol amendment 2, participants in the Double-blind Treatment Period discontinued all study interventions (islatravir [ISL], ulonivirine, or bictegravir/emtricitabine/tenofovir alafenamide [BIC/FTC/TAF]). Participants who received ISL + ulonivirine may have then entered the Unblinded Safety Monitoring Period and received standard of care non-study antiretroviral therapy (ART), provided by the investigator, until study completion or discontinuation.
Groups:
- Group 1: ISL 20 mg + Ulonivirine 100 mg: In the Double-blind Treatment Period, participants received ISL 20 mg + ulonivirine 100 mg once weekly (QW) and placebo to BIC/FTC/TAF once daily (QD). Following study-wide discontinuation of study intervention, participants may have entered the optional Unblinded Safety Monitoring Period and received standard of care non-study ART.
- Group 2: ISL 20 mg + Ulonivirine 200 mg: In the Double-blind Treatment Period, participants received ISL 20 mg + ulonivirine 200 mg QW and placebo to BIC/FTC/TAF QD. Following study-wide discontinuation of study intervention, participants may have entered the optional Unblinded Safety Monitoring Period and received standard of care non-study ART.
- Group 3: ISL 20 mg + Ulonivirine 400 mg: In the Double-blind Treatment Period, participants received ISL 20 mg + ulonivirine 400 mg QW and placebo to BIC/FTC/TAF QD. Following study-wide discontinuation of study intervention, participants may have entered the optional Unblinded Safety Monitoring Period and received standard of care non-study ART.
- Group 4: BIC/FTC/TAF: In the Double-blind Treatment Period, participants received placebo to ISL + placebo to ulonivirine QW and BIC/FTC/TAF 50 mg/200 mg/25 mg QD until study-wide discontinuation of study intervention.
Period: Double-blind Treatment Period
Arm/Group | Group 1: ISL 20 mg + Ulonivirine 100 mg | Group 2: ISL 20 mg + Ulonivirine 200 mg | Group 3: ISL 20 mg + Ulonivirine 400 mg | Group 4: BIC/FTC/TAF
Started | 40 | 41 | 40 | 40
Completed (Completed the Double-Blind Treatment Period as pre-specified in the protocol) | 37 | 39 | 38 | 39
Not Completed | 3 | 2 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 0
Period: Unblinded Safety Monitoring Period
Arm/Group | Group 1: ISL 20 mg + Ulonivirine 100 mg | Group 2: ISL 20 mg + Ulonivirine 200 mg | Group 3: ISL 20 mg + Ulonivirine 400 mg | Group 4: BIC/FTC/TAF
Started (Participants who entered the optional Unblinded Safety Monitoring Period) | 37 | 39 | 37 (Number started refers to only participants completing the Double-blind Treatment Period and volunteering to continue into the Unblinded Safety Monitoring Period) | 0 (The Unblinded Safety Monitoring Period was pre-specified in the protocol as available to participants in Groups 1, 2, and 3 only)
Completed | 25 | 25 | 24 | 0
Not Completed | 12 | 14 | 13 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 0
Not completed — Sponsor Decision | 5 | 6 | 4 | 0
Not completed — Withdrawal by Subject | 6 | 7 | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: ISL 20 mg + Ulonivirine 100 mg | Group 2: ISL 20 mg + Ulonivirine 200 mg | Group 3: ISL 20 mg + Ulonivirine 400 mg | Group 4: BIC/FTC/TAF | Total
Number analyzed (Participants) | 40 | 41 | 40 | 40 | 161
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.7 (12.1) | 46.5 (10.8) | 43.5 (12.6) | 47.9 (11.6) | 45.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 6 | 8 | 31
  Male | 31 | 33 | 34 | 32 | 130
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 6 | 8 | 28
  Not Hispanic or Latino | 30 | 30 | 32 | 32 | 124
  Unknown or Not Reported | 4 | 3 | 2 | 0 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 0 | 2
  Asian | 0 | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 14 | 13 | 13 | 50
  White | 27 | 24 | 27 | 26 | 104
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced One or More Adverse Events (AEs) During the Double-Blind Treatment Period +42 Days Post-Blind
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. As pre-specified in the protocol and supplemental statistical analysis plan (sSAP), presented here is the percentage of participants who experienced one or more AEs during the Double-blind Treatment Period and includes the 42 days following the final dose of double-blind study intervention.
Time Frame: Up to approximately 9 months
Population: All randomized participants who received at least 1 dose of double-blind study intervention
Measure: Number; unit: Percentage of Participants
Groups:
- Group 1: ISL 20 mg + Ulonivirine 100 mg: In the Double-blind Treatment Period, participants received ISL 20 mg + ulonivirine 100 mg QW and placebo to BIC/FTC/TAF QD.
- Group 2: ISL 20 mg + Ulonivirine 200 mg: In the Double-blind Treatment Period, participants received ISL 20 mg + ulonivirine 200 mg QW and placebo to BIC/FTC/TAF QD.
- Group 3: ISL 20 mg + Ulonivirine 400 mg: In the Double-blind Treatment Period, participants received ISL 20 mg + ulonivirine 400 mg QW and placebo to BIC/FTC/TAF QD.
- Group 4: BIC/FTC/TAF: In the Double-blind Treatment Period, participants received placebo to ISL + placebo to ulonivirine QW and BIC/FTC/TAF 50 mg/200 mg/25 mg QD.
Arm/Group | Group 1: ISL 20 mg + Ulonivirine 100 mg | Group 2: ISL 20 mg + Ulonivirine 200 mg | Group 3: ISL 20 mg + Ulonivirine 400 mg | Group 4: BIC/FTC/TAF
Number analyzed (Participants) | 40 | 41 | 40 | 40
Percentage of Participants | 75.0 | 75.6 | 80.0 | 67.5

2. Primary Outcome: Percentage of Participants Who Discontinued Study Intervention Due to an AE During the Double-Blind Treatment Period
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. As pre-specified in the protocol and sSAP, presented here is the percentage of participants who discontinued double-blind study intervention due to an AE during the Double-Blind Treatment Period.
Time Frame: Up to approximately 8 months
Population: All randomized participants who received at least 1 dose of double-blind study intervention
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: ISL 20 mg + Ulonivirine 100 mg | Group 2: ISL 20 mg + Ulonivirine 200 mg | Group 3: ISL 20 mg + Ulonivirine 400 mg | Group 4: BIC/FTC/TAF
Number analyzed (Participants) | 40 | 41 | 40 | 40
Percentage of Participants | 0.0 | 4.9 | 2.5 | 0.0

3. Primary Outcome: Percentage of Participants Who Experienced One or More AEs During the Unblinded Safety Monitoring Period
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. As pre-specified in the protocol and sSAP, presented here is the percentage of participants who experienced one or more AEs during the Unblinded Safety Monitoring Period, beginning 42 days following the final dose of double-blind study intervention.
Time Frame: Up to approximately 37 months
Population: All randomized participants who received at least 1 dose of double-blind study intervention and entered into the Unblinded Safety Monitoring Period
Measure: Number; unit: Percentage of Participants
Groups:
- Group 1: ISL 20 mg + Ulonivirine 100 mg: After receiving ISL 20 mg + ulonivirine 100 mg QW and placebo to BIC/FTC/TAF QD in the Double-blind Treatment Period, participants entered the Unblinded Safety Monitoring Period and received standard of care non-study ART.
- Group 2: ISL 20 mg + Ulonivirine 200 mg: After receiving ISL 20 mg + ulonivirine 200 mg QW and placebo to BIC/FTC/TAF QD in the Double-blind Treatment Period, participants entered the Unblinded Safety Monitoring Period and received standard of care non-study ART.
- Group 3: ISL 20 mg + Ulonivirine 400 mg: After receiving ISL 20 mg + ulonivirine 400 mg QW and placebo to BIC/FTC/TAF QD in the Double-blind Treatment Period, participants entered the Unblinded Safety Monitoring Period and received standard of care non-study ART.
Arm/Group | Group 1: ISL 20 mg + Ulonivirine 100 mg | Group 2: ISL 20 mg + Ulonivirine 200 mg | Group 3: ISL 20 mg + Ulonivirine 400 mg
Number analyzed (Participants) | 37 | 39 | 37
Percentage of Participants | 56.8 | 56.4 | 67.6

ADVERSE EVENTS:
Time Frame: Up to approximately 46 months (Double-blind Treatment Period: AEs were assessed at the participant level for up to approximately 9 months [from randomization to 42 days after last double-blind study intervention]; Unblinded Safety Monitoring Period: AEs were assessed at the participant level for up to approximately 37 months [beginning 42 days after the final double-blind study intervention to last participant data collection])
Description: All-Cause Mortality is reported for all randomized participants. Serious AEs and Other AEs are reported for all randomized participants who received at least 1 dose of study treatment. Double-blind Treatment Period arms include all events occurring up to 42 days following the final dose of double-blind study intervention. Unblinded Safety Monitoring Period arms include all events from 42 days after the final double-blind study intervention to study completion.
Groups:
- ISL 20 mg + MK-8507 100 mg QW: In the Double-blind Treatment Period, participants received ISL 20 mg + ulonivirine 100 mg once weekly (QW) and placebo to BIC/FTC/TAF once daily (QD).
- ISL 20 mg + MK-8507 200 mg QW: In the Double-blind Treatment Period, participants received ISL 20 mg + ulonivirine 200 mg QW and placebo to BIC/FTC/TAF QD.
- ISL 20 mg + MK-8507 400 mg QW: In the Double-blind Treatment Period, participants received ISL 20 mg + ulonivirine 400 mg QW and placebo to BIC/FTC/TAF QD.
- BIC/FTC/TAF QD: In the Double-blind Treatment Period, participants received placebo to ISL + placebo to ulonivirine QW and BIC/FTC/TAF 50 mg/200 mg/25 mg QD.
- ISL 20 mg + MK-8507 100 mg QW → Non-study ART: After receiving ISL 20 mg + ulonivirine 100 mg QW and placebo to BIC/FTC/TAF QD in the Double-blind Treatment Period, participants may have entered the optional Unblinded Safety Monitoring Period and received standard of care non-study ART.
- ISL 20 mg + MK-8507 200 mg QW → Non-study ART: After receiving ISL 20 mg + ulonivirine 200 mg QW and placebo to BIC/FTC/TAF QD in the Double-blind Treatment Period, participants may have entered the optional Unblinded Safety Monitoring Period and received standard of care non-study ART.
- ISL 20 mg + MK-8507 400 mg QW → Non-study ART: After receiving ISL 20 mg + ulonivirine 400 mg QW and placebo to BIC/FTC/TAF QD in the Double-blind Treatment Period, participants may have entered the optional Unblinded Safety Monitoring Period and received standard of care non-study ART.
Arm/Group | ISL 20 mg + MK-8507 100 mg QW | ISL 20 mg + MK-8507 200 mg QW | ISL 20 mg + MK-8507 400 mg QW | BIC/FTC/TAF QD | ISL 20 mg + MK-8507 100 mg QW → Non-study ART | ISL 20 mg + MK-8507 200 mg QW → Non-study ART | ISL 20 mg + MK-8507 400 mg QW → Non-study ART
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/41 | 0/40 | 0/40 | 0/37 | 0/39 | 0/37
Serious Adverse Events (participants affected / at risk) | 2/40 | 3/41 | 1/40 | 0/40 | 0/37 | 0/39 | 1/37
Other Adverse Events (participants affected / at risk) | 18/40 | 15/41 | 25/40 | 14/40 | 8/37 | 16/39 | 16/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ISL 20 mg + MK-8507 100 mg QW (N=40) | ISL 20 mg + MK-8507 200 mg QW (N=41) | ISL 20 mg + MK-8507 400 mg QW (N=40) | BIC/FTC/TAF QD (N=40) | ISL 20 mg + MK-8507 100 mg QW → Non-study ART (N=37) | ISL 20 mg + MK-8507 200 mg QW → Non-study ART (N=39) | ISL 20 mg + MK-8507 400 mg QW → Non-study ART (N=37)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related thrombosis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ISL 20 mg + MK-8507 100 mg QW (N=40) | ISL 20 mg + MK-8507 200 mg QW (N=41) | ISL 20 mg + MK-8507 400 mg QW (N=40) | BIC/FTC/TAF QD (N=40) | ISL 20 mg + MK-8507 100 mg QW → Non-study ART (N=37) | ISL 20 mg + MK-8507 200 mg QW → Non-study ART (N=39) | ISL 20 mg + MK-8507 400 mg QW → Non-study ART (N=37)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (4) | 6 (7) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (4) | 3 (3) | 5 (6) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 4 (4) | 7 (7) | 3 (3) | 4 (4) | 7 (7) | 11 (11)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (3) | 0 (0) | 2 (2) | 3 (4) | 1 (1) | 1 (1) | 1 (2)
Sinusitis (Infections and infestations) | 3 (4) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Syphilis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 4 (6) | 5 (10) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 5 (6) | 1 (1) | 4 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts and manuscripts regarding this trial prior to submission for publication. In accordance with standard editorial and ethical practice, the Sponsor will generally support publication of multi-center studies only in their entirety and not as individual site data. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (2):
  • Study Protocol (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT04564547/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-24): https://cdn.clinicaltrials.gov/large-docs/47/NCT04564547/SAP_001.pdf